CLINICAL TRIAL: NCT06176872
Title: Assessment of Cardiac CT Angiography in Patients Undergoing Thrombectomy for Ischemic Stroke
Brief Title: Cardiac CT Angiography in Patients With Acute Ischemic Stroke
Acronym: ACUTE
Status: Not yet recruiting | Type: Observational
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Collaborators: Siemens Healthcare Diagnostics Inc (Industry)
Responsible Party: Principal Investigator, Gabriel Broocks, Senior physician, Universitätsklinikum Hamburg-Eppendorf
Other Study IDs: 2022-100951-BO-ff
Record Dates: First submitted 2023-11-23; First posted 2023-12-20 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: Acute Ischemic Stroke; Coronary Artery Disease
Keywords: Computed Tomography Angiography
MeSH Terms: conditions — Ischemic Stroke; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cardiac Computed Tomography Angiography: Patients with acute ischemic stroke who receive cardiac computed tomography angiography as part of the routine diagnostic work-up of acute ischemic stroke.
  Interventions: Diagnostic Test: Cardiac Computed Tomography Angiography
- Retrospective matched cohort: A retrospective matched cohort of patients with acute ischemic stroke who did not receive cardiac computed tomography angiography.

INTERVENTIONS:
Diagnostic Test: Cardiac Computed Tomography Angiography — Non-invasive imaging of the heart, the greater vessels and the coronary arteries using computed tomography.
  Groups: Cardiac Computed Tomography Angiography

SUMMARY:
Mortality rates after acute ischemic stroke remain high despite continuously improving treatment. In this context, it is important to note that a relevant portion of acute ischemic stroke patients die from adverse cardiovascular events, such as myocardial infarction, rather than from complications associated with the stroke itself. A possible reason might be that this patient group often suffers from at least moderate asymptomatic coronary artery disease. This study seeks to integrate cardiac computed tomography angiography into the standard-of-care diagnostic protocol of acute ischemic stroke. The aim of this prospective mono-centric trial is to enable accurate diagnosis of therapy-relevant coronary artery disease, other concomitant cardiac findings and cardiac causes of acute ischemic stroke, without delaying stroke therapy. In the long-run, the goal is to investigate whether cardiac computed tomography angiography and the resulting therapeutic measures (interventions or medications added) can improve functional outcome and rate of adverse cardiac complications in patients with acute ischemic stroke compared to a retrospective matched-cohort of patients without cardiac CT imaging.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 40 years or above, presenting at the Emergency Department of the University Medical Center Hamburg-Eppendorf with a suspected acute ischemic stroke and a relevant neurological deficit (NIHSS score > 4).

Exclusion Criteria:

* A causal differential diagnosis for the acute stroke syndrome with absent intracranial vessel occlusion.
* No correlation for the patients' symptoms in the cranial CTA (no vessel obstruction).

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 40 years or above, presenting at the Emergency Department of the University Medical Center Hamburg-Eppendorf (primary care clinic) with a suspected AIS.
Sampling Method: Non-Probability Sample
Enrollment: 165 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2025-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Diagnosis of therapy-relevant CAD and concomitant cardiac findings resulting in new therapeutic measurements. | 1 day at hospital discharge
  Number of (newly) prescribed medications (e.g., anticoagulants), cardiac diagnostics/interventions/planned interventions, clinical status (NIHSS, mRs).

SECONDARY OUTCOMES:
The rate of adverse cardiovascular events (MACE). | 90 and 365 days
  rate of major adverse cardiovascular events (MACE).

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel Broocks, MD, Principal Investigator — Universitätsklinikum Hamburg-Eppendorf; Mathias Meyer, MD, Principal Investigator — Universitätsklinikum Hamburg-Eppendorf; Jennifer Erley, MD, Principal Investigator — Universitätsklinikum Hamburg-Eppendorf

IPD SHARING:
Plan to Share IPD: No
Due to data protection agreements, it is not possible to share the IPD. Nevertheless,parts of the datasets can be made available from the PIs upon reasonable request.